CLINICAL TRIAL: NCT06115239
Title: Evaluation of Changes in Quality of Life in Patients With Non-small Cell Lung Carcinoma Undergoing Lung Resection Before and After Receiving Adjuvant Treatment Using the EORTC-LC29 Questionnaire
Brief Title: QOL After SURGERY and ADJUVANT Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Pablo Fernandez Salvador, Principal Investigator, University of Salamanca
Other Study IDs: PI 2023 05 1296 - TD
Record Dates: First submitted 2023-10-16; First posted 2023-11-02 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Quality of Life
Keywords: Non-Small-Cell Lung Cancer; EORTC-LC29; Adjuvant Treatment; Pulmonary Resection; Quality of Life
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — The patients will fulfill the EORTC-LC29 and HADS questionnaires in 5 different moments.
  Other Names: Surveys

SUMMARY:
The goal of this prospective, observational study is to measure and analyze the effect of adjuvant treatment over the quality of life and recovery of patients undergoing pulmonary resection because of non-small cells lung cancer using the EORTC-LC29 questionnaire. The main question it aims to answer is:

Whether adjuvant systemic treatment affect or not the postoperative QOL of a NSCLC patient that underwent lung resection

Participants will fulfill two questionnaires (EORTC-LC29 and Hospital Anxiety and Depression Scale) in different stages of their treatment.

DETAILED DESCRIPTION:
Despite being surgery the preferred radical treatment of NSCLC in early stages, unforseen N2 disease, larger tumors or bad prognosis histological or molecular findings of the tumor will benefit of receiving adjuvant treatment.

As an adjuvant treatment, postoperative platinum-based chemotherapy has demonstrated its efficacy in increasing survival rates and reducing recurrence rates. Postoperative radiotherapy (RT) is limited due to decreased lung tolerance following surgery and conflicting results.

It is clear that lung cancer significantly impacts the quality of life of patients. According to the Lung Cancer Europe (LuCE) association, a survey conducted in 2021 with 515 patients revealed that 91.2% experienced limitations in their daily lives. Fatigue, sleep problems, cognitive difficulties, and significant reductions in physical activity were the main areas where patients reported the most complications. In addition to the inherent complications of cancer, we must consider the complications associated with surgery and systemic treatment.

Module LC29 is an update of the previous module published by the European Organisation for Research and Treatment of Cancer (EORTC), providing a more current perspective on lung cancer. This latest module retains 12 out of the 13 items from LC13 and adds 17 new items, which gather information on the side effects of medical and targeted therapies, as well as emotional problems. Furthermore, it includes 5 specific questions related to lung surgery. This multidisciplinary approach currently makes the LC29 questionnaire the most comprehensive tool for studying the quality of life of lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-85 years old
* Patients with any histological type of non-small-cell lung cancer in clinical stage T1C N0M0 or greater
* Patients that understand the purpose of the study, accept collaborate and sign the informed consent.

Exclusion Criteria:

* Patients not receiving adjuvant treatment due to complications, bad quality of life or express rejection at any moment of the curse of the process.
* Patients who cannot complete the previous questionnaires to assess their quality of life

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be formed by patients undergoing pulmonary resection because of lung cancer that are candidates of taking adjuvant treatment after surgery. The patients will be collected from the Thoracic Surgery Department of Hospital Clínico Universitario de Salamanca
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life before and after adjuvant treatment in patients undergoing pulmonary resection | Pre-surgery, seven days after surgery, before the first dose of adjuvant treatment, 2 days after the first dose of adjuvant treatment, 2 days after finishing the whole cycle of adjuvant treatment
  For quality of life assessment, patients will be asked to complete the Quality of Life Questionnaire Module LC29 (QLQ-LC29) of the European Organization for Research and Treatment of Cancer (EORTC).

SECONDARY OUTCOMES:
Correlation between the type of surgical procedure performed and postoperative quality of life | Before surgery, seven days after surgery
  Measure and analyze the correlation between the type of surgical procedure performed and postoperative quality of life upon completion of the surgical episode and before receiving any form of adjuvant treatment for lung cancer. Patients will be asked to complete the Quality of Life Questionnaire Module LC29 (QLQ-LC29) of the European Organization for Research and Treatment of Cancer (EORTC). The type of surgical procedure (segmentectomy, lobectomy or pneumonectomy), will be collected from the post-surgery report.
Correlation between the type of surgical approach performed and postoperative quality of life | Before surgery, seven days after surgery
  Measure and analyze the correlation between the type of surgical approach performed and postoperative quality of life upon completion of the surgical episode and before receiving any form of adjuvant treatment for lung cancer. Patients will be asked to complete the Quality of Life Questionnaire Module LC29 (QLQ-LC29) of the European Organization for Research and Treatment of Cancer (EORTC). The type of surgical approach (thoracotomy, VATS or RATS), will be collected from the post-surgery report.
Correlation between the occurrence of postoperative complications and a longer hospital stay | Before surgery, seven days after surgery, before the first dose of adjuvant treatment
  Analyze the correlation between the occurrence of postoperative complications and a longer hospital stay with the quality of life before receiving any form of adjuvant treatment for lung cancer. Patients will be asked to complete the Quality of Life Questionnaire Module LC29 (QLQ-LC29) of the European Organization for Research and Treatment of Cancer (EORTC). Post-surgery complications will be collected from the patient's medical record, recorded in the Jimena 4 software program. Hospital stay lenght will be collected from the patient´s hospital discharge report.
Effect of complications from adjuvant treatment on the surgical items of the EORTC-LC29 | Before the first dose of adjuvant treatment, 2 days after the first dose of adjuvant treatment, 2 days after finishing the whole cycle of adjuvant treatment
  Measure and analyze the effect of complications from adjuvant treatment on the surgical items of the EORTC-LC29 for patients undergoing lung resection for lung cancer. Patients will be asked to complete the Quality of Life Questionnaire Module LC29 (QLQ-LC29) of the European Organization for Research and Treatment of Cancer (EORTC), where higher score represents higher level of symptomatology or problems.
Adjuvant chemotherapy/immunotherapy treatment regimen significantly decreases the quality of life | Before the first cycle of adjuvant treatment, 2 days after the first dose of adjuvant treatment, 2 days after finishing the whole cycle of adjuvant treatment
  Measure and analyze whether any adjuvant chemotherapy/immunotherapy treatment regimen significantly decreases the quality of life of patients who receive adjuvant treatment after undergoing lung resection compared to others.
Correlation between the presence of Chronic Obstructive Pulmonary Disease (COPD) and postoperative quality of life | Before surgery, seven days after surgery, before the first dose of adjuvant treatment, 2 days after the first dose of adjuvant treatment, 2 days after finishing the whole cycle of adjuvant treatment
  Analyze the correlation between the presence of Chronic Obstructive Pulmonary Disease (COPD) and postoperative quality of life upon completion of the surgical episode before and after receiving any form of adjuvant treatment for lung cancer. Patients will be asked to complete the Quality of Life Questionnaire Module LC29 (QLQ-LC29) of the European Organization for Research and Treatment of Cancer (EORTC).
Level of anxiety/depression in patients undergoing lung resection before and after receiving the first cycle of adjuvant treatment | Before the first dose of adjuvant treatment, 2 days after the first dose of adjuvant treatment, 2 days after finishing the whole cycle of adjuvant treatment
  Measure and analyze the level of anxiety/depression in patients undergoing lung resection before and after receiving the first cycle of adjuvant treatment for lung cancer. Patients will be asked to complete the HADS questionnaire.
Effect of Performance Status (PS) and pre-adjuvant treatment ECOG on the quality of life after receiving the first cycle of any treatment modality. | Before the first dose of adjuvant treatment, 2 days after the first dose of adjuvant treatment, 2 days after finishing the whole cycle of adjuvant treatment
  Measure and analyze the effect of Performance Status (PS) and pre-adjuvant treatment ECOG on the quality of life after receiving the first cycle of any treatment modality. Patients will be asked to complete the Quality of Life Questionnaire Module LC29 (QLQ-LC29) of the European Organization for Research and Treatment of Cancer (EORTC). Performance Status Score and ECOG score data will be collected from the patient's medical record, recorded in the Jimena 4 software program.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Fernández Salvador, Nurse, Principal Investigator — University of Salamanca; Nuria M Novoa Valentín, MD, PhD, Study Director — University of Salamanca; Marta G Fuentes Gago, MD, PhD, Study Director — University of Salamanca; María B García Cenador, MD, PhD, Study Chair — University of Salamanca
Locations (1):
- Hospital Clínico Universitario, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: After recruitment has finalized

REFERENCES:
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Nicholson AG, Tsao MS, Beasley MB, Borczuk AC, Brambilla E, Cooper WA, Dacic S, Jain D, Kerr KM, Lantuejoul S, Noguchi M, Papotti M, Rekhtman N, Scagliotti G, van Schil P, Sholl L, Yatabe Y, Yoshida A, Travis WD. The 2021 WHO Classification of Lung Tumors: Impact of Advances Since 2015. J Thorac Oncol. 2022 Mar;17(3):362-387. doi: 10.1016/j.jtho.2021.11.003. Epub 2021 Nov 20. PMID 34808341
- [Background] Ettinger DS, Wood DE, Aisner DL, Akerley W, Bauman JR, Bharat A, Bruno DS, Chang JY, Chirieac LR, D'Amico TA, DeCamp M, Dilling TJ, Dowell J, Gettinger S, Grotz TE, Gubens MA, Hegde A, Lackner RP, Lanuti M, Lin J, Loo BW, Lovly CM, Maldonado F, Massarelli E, Morgensztern D, Ng T, Otterson GA, Pacheco JM, Patel SP, Riely GJ, Riess J, Schild SE, Shapiro TA, Singh AP, Stevenson J, Tam A, Tanvetyanon T, Yanagawa J, Yang SC, Yau E, Gregory K, Hughes M. Non-Small Cell Lung Cancer, Version 3.2022, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2022 May;20(5):497-530. doi: 10.6004/jnccn.2022.0025. PMID 35545176
- [Background] Shi Y, Wu S, Ma S, Lyu Y, Xu H, Deng L, Chen X. Comparison Between Wedge Resection and Lobectomy/Segmentectomy for Early-Stage Non-small Cell Lung Cancer: A Bayesian Meta-analysis and Systematic Review. Ann Surg Oncol. 2022 Mar;29(3):1868-1879. doi: 10.1245/s10434-021-10857-7. Epub 2021 Oct 6. PMID 34613537
- [Background] Atkins BZ, Harpole DH Jr, Mangum JH, Toloza EM, D'Amico TA, Burfeind WR Jr. Pulmonary segmentectomy by thoracotomy or thoracoscopy: reduced hospital length of stay with a minimally-invasive approach. Ann Thorac Surg. 2007 Oct;84(4):1107-12; discussion 1112-3. doi: 10.1016/j.athoracsur.2007.05.013. PMID 17888955
- [Background] Scott WJ, Allen MS, Darling G, Meyers B, Decker PA, Putnam JB, McKenna RW, Landrenau RJ, Jones DR, Inculet RI, Malthaner RA. Video-assisted thoracic surgery versus open lobectomy for lung cancer: a secondary analysis of data from the American College of Surgeons Oncology Group Z0030 randomized clinical trial. J Thorac Cardiovasc Surg. 2010 Apr;139(4):976-81; discussion 981-3. doi: 10.1016/j.jtcvs.2009.11.059. Epub 2010 Feb 20. PMID 20172539
- [Background] Whitson BA, Groth SS, Duval SJ, Swanson SJ, Maddaus MA. Surgery for early-stage non-small cell lung cancer: a systematic review of the video-assisted thoracoscopic surgery versus thoracotomy approaches to lobectomy. Ann Thorac Surg. 2008 Dec;86(6):2008-16; discussion 2016-8. doi: 10.1016/j.athoracsur.2008.07.009. PMID 19022040
- [Background] Pignon JP, Tribodet H, Scagliotti GV, Douillard JY, Shepherd FA, Stephens RJ, Dunant A, Torri V, Rosell R, Seymour L, Spiro SG, Rolland E, Fossati R, Aubert D, Ding K, Waller D, Le Chevalier T; LACE Collaborative Group. Lung adjuvant cisplatin evaluation: a pooled analysis by the LACE Collaborative Group. J Clin Oncol. 2008 Jul 20;26(21):3552-9. doi: 10.1200/JCO.2007.13.9030. Epub 2008 May 27. PMID 18506026
- [Background] Butts CA, Ding K, Seymour L, Twumasi-Ankrah P, Graham B, Gandara D, Johnson DH, Kesler KA, Green M, Vincent M, Cormier Y, Goss G, Findlay B, Johnston M, Tsao MS, Shepherd FA. Randomized phase III trial of vinorelbine plus cisplatin compared with observation in completely resected stage IB and II non-small-cell lung cancer: updated survival analysis of JBR-10. J Clin Oncol. 2010 Jan 1;28(1):29-34. doi: 10.1200/JCO.2009.24.0333. Epub 2009 Nov 23. PMID 19933915
- [Background] Wang SF, Mao NQ, Zhao WH, Pan XB. Postoperative radiotherapy in pIIIA-N2 non-small cell lung cancer after complete resection and adjuvant chemotherapy: A meta-analysis. Medicine (Baltimore). 2022 Jul 15;101(28):e29550. doi: 10.1097/MD.0000000000029550. PMID 35839025
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Shukla N, Hanna N. Neoadjuvant and Adjuvant Immunotherapy in Early-Stage Non-Small Cell Lung Cancer. Lung Cancer (Auckl). 2021 Jun 28;12:51-60. doi: 10.2147/LCTT.S277717. eCollection 2021. PMID 34234606
- [Background] Broderick SR. Adjuvant and Neoadjuvant Immunotherapy in Non-small Cell Lung Cancer. Thorac Surg Clin. 2020 May;30(2):215-220. doi: 10.1016/j.thorsurg.2020.01.001. PMID 32327180
- [Background] Paz-Ares L, Luft A, Vicente D, Tafreshi A, Gumus M, Mazieres J, Hermes B, Cay Senler F, Csoszi T, Fulop A, Rodriguez-Cid J, Wilson J, Sugawara S, Kato T, Lee KH, Cheng Y, Novello S, Halmos B, Li X, Lubiniecki GM, Piperdi B, Kowalski DM; KEYNOTE-407 Investigators. Pembrolizumab plus Chemotherapy for Squamous Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Nov 22;379(21):2040-2051. doi: 10.1056/NEJMoa1810865. Epub 2018 Sep 25. PMID 30280635
- [Background] Gabay C, Russo A, Raez LE, Rolfo Cervetto C. Adjuvant therapy in non-small cell lung cancer: is targeted therapy joining the standard of care? Expert Rev Anticancer Ther. 2021 Nov;21(11):1229-1235. doi: 10.1080/14737140.2021.1982387. Epub 2021 Sep 25. PMID 34528869
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Pompili C. Quality of life after lung resection for lung cancer. J Thorac Dis. 2015 Apr;7(Suppl 2):S138-44. doi: 10.3978/j.issn.2072-1439.2015.04.40. PMID 25984359
- [Background] Koller M, Warncke S, Hjermstad MJ, Arraras J, Pompili C, Harle A, Johnson CD, Chie WC, Schulz C, Zeman F, van Meerbeeck JP, Kulis D, Bottomley A; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Group; EORTC Lung Cancer Group. Use of the lung cancer-specific Quality of Life Questionnaire EORTC QLQ-LC13 in clinical trials: A systematic review of the literature 20 years after its development. Cancer. 2015 Dec 15;121(24):4300-23. doi: 10.1002/cncr.29682. Epub 2015 Oct 9. PMID 26451520
- [Background] Koller M, Hjermstad MJ, Tomaszewski KA, Tomaszewska IM, Hornslien K, Harle A, Arraras JI, Morag O, Pompili C, Ioannidis G, Georgiou M, Navarra C, Chie WC, Johnson CD, Himpel A, Schulz C, Bohrer T, Janssens A, Kulis D, Bottomley A. An international study to revise the EORTC questionnaire for assessing quality of life in lung cancer patients. Ann Oncol. 2017 Nov 1;28(11):2874-2881. doi: 10.1093/annonc/mdx453. PMID 28945875
- [Background] Pompili C, Koller M, Velikova G. Choosing the right survey: the lung cancer surgery. J Thorac Dis. 2020 Nov;12(11):6892-6901. doi: 10.21037/jtd.2019.12.131. PMID 33282392
- See also: 6th LuCE Report on lung cancer. Experiences and quality of life of people impacted by lung cancer in Europe — https://www.lungcancereurope.eu/wp-content/uploads/2022/06/6th-LuCE-Report_Web-version_Definitive.pdf